CLINICAL TRIAL: NCT01690026
Title: Facilitating Adolescent Self-Change for Alcohol Problems
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Diego (Other)
Responsible Party: Principal Investigator, Sandra Brown, Vice-Chancellor of Research, University of California, San Diego
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Treatment
Other Study IDs: Project Options
Record Dates: First submitted 2012-09-12; First posted 2012-09-21 (Estimated); Last update posted 2017-11-06 (Actual); Status verified 2017-11

CONDITIONS: Underage Drinking
MeSH Terms: conditions — Underage Drinking

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Brief intervention (Other): Motivational intervention based brief intervention
  Interventions: Behavioral: Motivation interviewing based brief intervention
- Standard intervention (Other): Standard intervention condition
  Interventions: Behavioral: Standard Intervention

INTERVENTIONS:
Behavioral: Motivation interviewing based brief intervention
  Arms: Brief intervention
Behavioral: Standard Intervention
  Arms: Standard intervention

SUMMARY:
This present multi-site investigation compares a voluntary brief intervention for adolescent alcohol problems to an educational comparison condition. Measures are taken at intake and at 4 and 12 weeks post intake to determine effectiveness of the intervention to promote personal change efforts and arrest progression of alcohol problems. This study tests cognitive mechanisms of change and treatment characteristics and processes associated with youth self-regulation to reduce or stop hazardous drinking.

ELIGIBILITY:
Inclusion Criteria:

* All 9th-12th graders at six schools from 3 sites across the country are eligible to participate, regardless of alcohol experience

Exclusion Criteria:

* exclusion prior to 9th grade and after 12th grade

Ages: 14 Years to 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 1209 (Actual)
Dates: Start 2012-10; Primary Completion 2017-03 (Actual); Study Completion 2017-06-30 (Actual)

PRIMARY OUTCOMES:
Alcohol use and problems | one year

SECONDARY OUTCOMES:
Cognitive mediators | one year

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - Drug Free Youth in Town, Miami, Florida
  - University of Minnesota, Minneapolis, Minnesota
  - Reed College, Portland, Oregon